CLINICAL TRIAL: NCT01063504
Title: Teriparatide for Improved Knee Prosthesis Fixation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Per Aspenberg, professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PTHKnee
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teriparatide 20 microgram daily for 2 months (Active Comparator)
  Interventions: Drug: teriparatide
- Placebo (Placebo Comparator)
  Interventions: Drug: teriparatide

INTERVENTIONS:
Drug: teriparatide

SUMMARY:
The investigators will study how well knee joint prostheses become fixed to the bone when patients get teriparatide, compared to placebo. Measurements will use high resolution 3D radiography (radiostereometry, RSA).

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee planned for prosthesis surgery

Exclusion Criteria:

* Poor health, drugs affecting bone metabolism.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Migration as measured by RSA maximal total point motion. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Motala hospital, Motala, Sweden